CLINICAL TRIAL: NCT05346575
Title: Teaching Obesity Treatment Options to Adult Learners (TOTAL): A Multi-site RCT
Brief Title: TOTAL: A Multisite RCT
Acronym: TOTAL
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: IIR 20-322; 2021-1441 (Other: UW IRB)
Record Dates: First submitted 2022-04-18; First posted 2022-04-26 (Actual); Last update posted 2025-10-27 (Actual); Status verified 2025-10

CONDITIONS: Obesity; Overweight
Keywords: Bariatric Surgery; Weight-Loss Drugs; Diet, Therapy; Physical Activity; Body Mass Index; Veteran
MeSH Terms: conditions — Obesity; Overweight; Motor Activity

STUDY DESIGN:
Intervention Model Description: A multi-site, two-arm, parallel randomized control trial to test the effectiveness of the TOTAL intervention vs. usual care on initiation if obesity treatment among Veterans with overweight/obesity.
Who Masked: Investigator, Outcomes Assessor
Masking Description: All study team members will be blinded to the block randomization sizes except the biostatisticians. Outcome assessors will be masked to a participants randomization assignment. Interventionists (Study team member administering the TOTAL intervention) will notify participants randomized to the TOTAL intervention. The outcomes assessor will administer assessment surveys to all participants and will remain blinded from each participants intervention status.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Usual Care (Active Comparator): Participants randomized to this arm will receive the usual obesity care, but will complete assessments every 6 months.
  Interventions: Behavioral: Usual care
- TOTAL intervention (Experimental): Participants randomized to this arm will watch the TOTAL intervention video and participate in 1:1 motivational sessions every 6 months. Participants will also complete assessments every 6 months.
  Interventions: Behavioral: Teaching Obesity Treatments to Adult Learners (TOTAL)

INTERVENTIONS:
Behavioral: Teaching Obesity Treatments to Adult Learners (TOTAL) — TOTAL includes both video component and motivational telemedicine calls delivered via VA Video Connect (VVC) by a study interventionist. We will invite study participants to watch the 18-minute video at least once. The motivational component of TOTAL will consist of three telemedicine-based (VVC), one-on-one, 30-minute calls at 1 week, 6 months, and 12 months after randomization. This timing was selected so Veterans would have regular interactions with the interventionist within one year of initiating the intervention. Each motivational session will be tailored to where Veterans are in the treatment initiation process. Electronic outcome assessment surveys will be sent to the participants at baseline, at each motivational telemedicine visit, and for the 18 month assessment.
  Arms: TOTAL intervention
Behavioral: Usual care — The usual care group will be electronically sent the 1-week, 6-month, 12-month, 18-month assessments. All usual care participants will be offered the opportunity to watch the educational video component of TOTAL after the final outcome assessment is performed (18 months post-randomization). Veterans in the usual care arm will also have access to the MOVE! program via referrals from the PCP or self-referral to MOVE!. If they initiate treatment in MOVE!, they may progress through MOVE! and receive obesity medications or be referred for bariatric surgery if they choose to do so.
  Arms: Usual Care

SUMMARY:
Nearly 8 in 10 Veterans meet criteria for overweight/obesity. Three evidence-based treatment options are available within VA (behavioral weight management [MOVE!], obesity medications, and bariatric surgery).

However, all treatments are significantly underutilized. This study will evaluate the effectiveness of a novel intervention designed to increase obesity treatment initiation and subsequently weight loss within VA. The intervention, Teaching Obesity Treatment Options to Adult Learners (TOTAL), involves an educational video and multiple motivational sessions delivered via telemedicine. If effective, TOTAL could be implemented throughout VA without requiring significant resources and could be integrated into the existing VA behavioral weight management program, MOVE!, which is present at nearly every VA medical center.

DETAILED DESCRIPTION:
Background: Nearly 80% of Veterans meet criteria for overweight (body mass index [BMI] of 25-29.9 kg/m2) or obesity (BMI 30). VA offers three evidence-based obesity treatments at little to no cost to Veterans: MOVE! (to improve dietary intake and physical activity through behavioral modification); obesity medications; and bariatric surgery, but all are significantly underutilized: <10% of Veterans with obesity participate in MOVE!; 2% receive obesity medications; and 0.3% of those who meet BMI criteria for bariatric surgery (BMI 35) undergo it. There is an urgent need to increase use of all three treatments to improve Veteran health.

Significance/Impact: Nearly 4,000,000 Veterans meet BMI criteria for overweight/obesity. It is essential that Veterans with overweight/obesity are aware of the three treatment options and are motivated to pursue them. Currently, no interventions in VA seek to increase use of all three evidence-based obesity treatment options for Veterans not currently participating in MOVE!. The TOTAL intervention (Teaching Obesity Treatment Options to Adults Learners), if effective, would increase obesity treatment initiation for Veterans, lead to greater weight loss, and improve quality of life. Given that TOTAL is deliverable via VA telemedicine, it could be implemented throughout the VA healthcare system without requiring significant resources and could be integrated into the existing VA behavioral weight management program, MOVE!.

Innovation: The research in this proposal would be the first adequately powered RCT in VA testing an intervention to increase use of all three evidence-based obesity treatments: MOVE!, obesity medications, and bariatric surgery. It would leverage the power of the VA electronic health record and would improve access to care by expanding use of a recently developed telemedicine technology - VA Video Connect (VVC) - which was developed by VA researchers. It could be implemented and disseminated efficiently within VA given that MOVE! is available at every VAMC and is supported by NCP.

Specific Aims: Aim 1: Compare the effectiveness of TOTAL vs. usual care for increasing obesity treatment initiation among Veterans with overweight/obesity who are not participating in MOVE!; Aim 2: Compare the effectiveness of TOTAL vs. usual care for increasing sustained MOVE! participation, receipt of an obesity medication prescription or bariatric surgery referral, and weight loss; Aim 3: Inform future dissemination efforts of TOTAL via interviews with key stakeholders, a "Reach" analysis, and cost analysis.

Methodology: Study population: Veterans at two VAMCs, age 18-75 with a BMI 30 or 27-29.9 + an obesity related comorbidity who have not had a MOVE! visit within the past 12 months and thus are not participating in obesity treatment will participate in the RCT; Intervention: The TOTAL intervention consists of an 18-minute obesity treatment educational video and three motivational sessions (all delivered via VA Video Connect [VVC]); Comparison: Usual care (Veterans who have not had a MOVE! visit in the previous 12 months); Outcomes: MOVE! initiation, sustained MOVE! participation, obesity medication use, bariatric surgery referral, weight change; Timing: Primary and secondary outcomes will be measured 18 months post-randomization.

Implementation/Next Steps: Facilitators and barriers to TOTAL implementation will be assessed in Aim 3 interviews with Veteran, provider, and operations stakeholders using the Consolidated Framework for Implementation Research (CFIR). The investigators will also perform "reach" and cost analyses. The investigators will collaborate with NCP to disseminate TOTAL to all VAMCs that have a MOVE! program. The National MOVE! Director will present study results on a national MOVE! call and make presentation materials available on the national MOVE! SharePoint dissemination site. The National MOVE! Director will support MOVE! coordinators who work directly with health behavior coordinators at every VAMC with MOVE!. The study team will consider partnering with NCP to conduct a QUERI National Partnered Evaluation evaluating how TOTAL can be implemented throughout VA.

ELIGIBILITY:
Inclusion Criteria:

* Veterans will be eligible for this study if they have had no MOVE! visit attendance within the last 12 months, no previous bariatric surgery, not currently on weight loss medications, and a BMI of 30 kg/m2 or 27-29.9 + an obesity-related comorbidity

Exclusion Criteria:

* Veterans will be not be eligible for this study if they are pregnant or are planning to become pregnant within the study period, currently breast feeding, have cancer not in remission, do not have access to a telephone, have severe hearing/visual impairment, weigh more than 420 lbs (due to scale limitations).

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 440 (Actual)
Dates: Start 2023-01-23 (Actual); Primary Completion 2026-08-31 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Obesity treatment initiation | 18 months
  Attendance at an individual or group MOVE! visit within 18 months of randomization. Assessed at baseline and 18 months via VA electronic health record review.

SECONDARY OUTCOMES:
Sustained obesity treatment | 18 months
  Attendance at 12 or more MOVE! visits (individual or group) over 18 months. Assessed via VA electronic health record review at baseline and 18 months.
Obesity medication initiation | 18 months
  Presence of an obesity medication on the active medications list within the VA electronic health record. Assessed at baseline and 18months
Bariatric surgery referral | 18 months
  Receipt of a bariatric surgery referral. Assessed at baseline and 18 months via VA electronic health record review.
Weight Change | 18 months
  Patient will weigh themselves on a calibrated scale provided by the study. Patients will enter their weight in an electronic survey sent to them every 6 months (baseline, 6 months, 12months, and 18 months). Participants will also send a picture of their weight on the scale to verify the number.

CONTACTS AND LOCATIONS:
Overall Officials: Luke M Funk, MD MPH, Principal Investigator — William S. Middleton Memorial Veterans Hospital, Madison, WI
Locations (2):
- United States (2):
  - VA Greater Los Angeles Healthcare System, West Los Angeles, CA, West Los Angeles, California
  - William S. Middleton Memorial Veterans Hospital, Madison, WI, Madison, Wisconsin

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2023-04-13): https://cdn.clinicaltrials.gov/large-docs/75/NCT05346575/ICF_000.pdf